CLINICAL TRIAL: NCT06960421
Title: An eXercise-based Frailty Intervention in Lung Transplantation (XFIT): A Phase Ib Clinical Trial Focused on Establishing Safety
Brief Title: Exercise-based Frailty Intervention in Lung Transplantation (XFIT)
Acronym: XFIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Pennsylvania (Other); University of North Carolina (Other); Columbia University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25-43803; 1R61HL169183 (NIH)
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Frailty; Lung Tranplant Candidate
Keywords: frailty; lung transplant; prehabilitation; remote intervention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: We will randomize 1:1 into XFIT intervention versus enhanced standard of care using sex and frailty severity as stratification variables
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XFIT (Active Comparator): XFIT is an 8-week telehealth-delivered, home-based exercise/behavior modification intervention. It integrates theoretical frameworks of behavior change to engage frail lung transplant candidates in program of pre-habilitation.
  Interventions: Behavioral: XFIT
- Enhanced standard of care (No Intervention): Participants in ESC will be provided with individualized recommendations to improve physical frailty tailored to their baseline assessments, as well as contemporary information on treatments for physical frailty published by the NIH's Science of Frailty group (https://frailtyscience.org/). ESC participants will not engage in weekly treatment sessions, wear activity trackers throughout the intervention period, or receive the personalized psychological treatment provided to those in XFIT.

INTERVENTIONS:
Behavioral: XFIT — XFIT is an 8-week telehealth-delivered, home-based exercise/behavior modification intervention. It integrates theoretical frameworks of behavior change to engage frail lung transplant candidates in program of pre-habilitation.
  Arms: XFIT

SUMMARY:
The goal of XFIT study is to measure the safety of an 8-week telehealth-delivered exercise and behavioral training program to treat frailty in lung transplant candidates in their own home. The main questions XFIT aims to answer are:

* Is XFIT safe?
* Is XFIT feasible and acceptable by participants?
* Is XFIT effective in improving frailty and physical function as reflected in patient-reported outcomes.

Participants will:

- Participate in the 8-week XFIT program or enhanced standard of care

DETAILED DESCRIPTION:
We will randomize 70 patients who reflect the diversity and spectrum of illness seen in the general lung transplant candidate population to either XFIT or enhanced standard of care. An interventionalist with expertise in exercise physiology and remote interventions will deliver 8 weekly sessions using video-conference software in participants' homes. These sessions feature one-on-one exercise training and targeting of behavioral barriers to optimizing physical activity using motivational interviewing principles. Establishing safety is our primary outcome. We will secondarily establish feasibility and acceptability, and explore responsiveness six-minute walk distance, frailty, Patient Reported Outcomes . We anticipate that this first-of-its kind study in solid organ transplantation will establish fundamental safety, feasibility, and accessibility data needed inform larger scale interventions.

ELIGIBILITY:
Group 1

Inclusion Criteria:

* Age 18 - 65 years
* Lung Transplant Candidates
* Speaks English or Spanish
* ≤ 8LPM O2 on 6MWT
* SPPB score ≤ 10

Exclusion Criteria:

* Lives Alone
* BMI < 18.0 kg/m2
* Engaged in clinical pulmonary rehabilitation program
* Severe pHTN (RHC mPAP ≥ 30 mmHg or TTE PASP ≥ 60mmHg or moderately/severely reduced RV systolic function on TTE
* Deemed unsafe by site PI

Group 2

Inclusion Criteria:

* Age 18 - 75 years
* Speaks English or Spanish
* ≤ 15LPM O2 on 6MWT
* SPPB score ≤ 10

Exclusion Criteria:

* Lives Alone
* BMI < 18.0 kg/m2
* Engaged in clinical pulmonary rehabilitation program
* Severely reduced RV systolic function on TTE
* Deemed unsafe by site PI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-07-15 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Death | 8 weeks
Major cardiovascular event | 8 weeks
> 2 unplanned hospitalizations | 8 weeks

SECONDARY OUTCOMES:
Desaturation | 8 weeks
Coughing | 8 weeks
Presyncope | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Singer, MD, MS, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California,San Francisco, San Francisco, California
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
An anonymized dataset with key study-related data will be made available to investigators upon request one-year after the publication of the primary study findings. Investigators will be able to make requests through Drs. Singer and Smith, who can facilitate such data management tasks. In addition, we will plan to provide a complete, anonymized dataset for deposition into online data repositories within three years of publication of our primary findings, for use in subsequent follow-up analyses or meta-analytic studies. We will also make annotated statistical analytical code available for public usage, in order to increase reproducibility of findings for future studies. We will also make available our final protocol. These data will be available in an online data repository for as long as the repository is able to host them. They will also be available for request from Drs. Singer and Smith.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As detailed above. The trial is expected to run from July 2026 to June 2029.
Access Criteria: As above.

REFERENCES:
- See also: NIH Reporter study description — https://reporter.nih.gov/search/XKBKrqavSEC54l_xwGXt-A/project-details/10952296